CLINICAL TRIAL: NCT05009784
Title: Effects of Natural Sounds on Attention Restoration in Noisy Environment
Acronym: EARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanyang Technological University (Other)
Collaborators: National Research Foundation, Singapore (Other Government); Ministry of National Development, Singapore (Other Government); Housing and Development Board, Singapore (Other Government)
Responsible Party: Principal Investigator, Georgios CHRISTOPOULOS, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COT-V4-2020-1-S001
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cognitive Fatigue; Mental Fatigue; Heart Rate Variability; Skin Conductance; Behavioral Performance; Positive and Negative Affect; Inhibition; Working Memory; Perceived Restoration
MeSH Terms: conditions — Mental Fatigue; Inhibition, Psychological | interventions — BaseLine dental cement; SIR1 protein, S cerevisiae

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traffic Sound (Active Comparator): 600 seconds of traffic sound
  Interventions: Other: Baseline; Other: Fatigue Manipulation; Other: Traffic Sound
- Traffic and Masking Sounds (Experimental): 600 seconds of traffic and masking sound
  Interventions: Other: Baseline; Other: Fatigue Manipulation; Other: Traffic and Masking Sound
- Silence (Active Comparator): 600 seconds of no sound
  Interventions: Other: Baseline; Other: Fatigue Manipulation; Other: Silence

INTERVENTIONS:
Other: Baseline — 5-min urban park video clip (Presented on a TV)
Other: Fatigue Manipulation — 20-min 2-back task (Presented on a computer)
Other: Traffic Sound — Active Comparator: Traffic Sound (Played through speakers)
  Arms: Traffic Sound
Other: Traffic and Masking Sound — Experimental: Traffic and Masking Sound (Played through speakers)
  Arms: Traffic and Masking Sounds
Other: Silence — No Intervention: No sound (Played through speakers)
  Arms: Silence

SUMMARY:
This study aims to examine whether listening to natural sounds in a noisy (traffic) environment compared to traffic noise only impacts behavioural, cognitive, affective, and physiological markers associated with attention restoration. Attention restoration will be examined as an aspect of cognitive fatigue.

DETAILED DESCRIPTION:
Based on the Attention Restoration Theory (Kaplan, 1995), we hypothesize that listening to natural sounds has restorative effects on attention by supporting greater use of involuntary attention. This generates the prediction that exposure to natural sounds in the context of a noisy environment will have greater restorative effects on attention (i.e., physiological, affect, cognition, and behaviour) as compared to the control group (exposed to noise only). Individual differences (i.e., age, gender, caffeine and food intake, body mass index, skin temperature, noise sensitivity, sleep quality, baseline physiology and behavioural performance) will be examined and accounted for. A cognitive task will be administered at the beginning of the experiment to induce fatigue to examine the restorative effects of natural sounds.

ELIGIBILITY:
Inclusion Criteria:

* Singapore-based
* Non-clinical
* 18-35years

Exclusion Criteria:

* Individuals with hearing difficulties or failing to meet the minimal threshold for normal hearing
* Individuals with a history of ear, developmental, neurological, or psychiatric disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 162 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Reverse Corsi Task (Change) | up to 1 hour before and after sound intervention
  Change in Span
Reverse Corsi Task (Change) | up to 1 hour before and after sound intervention
  Change in Reaction Time
Go/NoGo Task (Change) | up to 1 hour before and after sound intervention
  Change in Accuracy
Go/NoGo Task (Change) | up to 1 hour before and after sound Intervention
  Change in Reaction Time
Electrocardiograph (Change) | up to 1 hour before and after sound intervention
  Change in Heart Rate Variability
Electrodermal Activity (Change) | up to 1 hour before and after sound intervention
  Change in Skin Conductance Level
Electrodermal Activity (Change) | up to 1 hour before and after sound intervention
  Change in Skin Conductance Response
Positive and Negative Affect Schedule - Expanded Form (Change) | up to 1 hour before and after sound intervention
  Change in Positive Affect Score
Positive and Negative Affect Schedule - Expanded Form (Change) | up to 1 hour before and after sound intervention
  Change in Negative Affect Score
Fatigue State Questionnaire (Change) | up to 1 hour before and after sound intervention
  Change in Fatigue State Questionnaire Score

SECONDARY OUTCOMES:
Perceived Restorativeness Soundscape Scale | up to 1 hour after sound Intervention
  Perceived Restorativeness Soundscape Scale Score

CONTACTS AND LOCATIONS:
Locations (1):
- Cultural Science Innovations, Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarsson JJ, Wiens S, Nilsson ME. Stress recovery during exposure to nature sound and environmental noise. Int J Environ Res Public Health. 2010 Mar;7(3):1036-46. doi: 10.3390/ijerph7031036. Epub 2010 Mar 11. PMID 20617017
- [Background] Kaplan S. The restorative benefits of nature: Toward an integrative framework. J. Environ. Psychol. 1995; 15(3): 169-182.